CLINICAL TRIAL: NCT01365195
Title: Intraoperative Ketamine Administration in Colorectal Surgery: Effect on Postoperative Clinical Outcomes
Brief Title: Effect of Ketamine on Postoperative Clinical Outcomes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment failure
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00024533
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Surgery
Keywords: opioid; Fentanyl; Anesthetic adjuvant; Pain management; Perioperative outcomes; Constipation; Ileus; Colorectal
MeSH Terms: conditions — Agnosia; Constipation; Ileus | interventions — Saline Solution; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Loading and Infusion:
  Saline at infusion rate calculated and adjusted for weight to match ketamine bolus-infusion rate
  Interventions: Drug: Ketamine high-dose; Drug: Ketamine low-dose
- Ketamine low-dose (Active Comparator): Loading: 0.5 mg/Kg Infusion: 5 mcg/kg/min
  Interventions: Drug: Placebo; Drug: Ketamine high-dose
- Ketamine high-dose (Active Comparator): Loading: 1 mg/Kg Infusion: 10 mcg/kg/min
  Interventions: Drug: Placebo; Drug: Ketamine low-dose

INTERVENTIONS:
Drug: Placebo — Loading and Infusion: Saline at infusion rate calculated and adjusted for weight to match ketamine bolus-infusion rate
  Other Names: Saline Solution
  Arms: Ketamine high-dose; Ketamine low-dose
Drug: Ketamine high-dose — Loading: 1 mg/Kg Infusion: 10 mcg/kg/min
  Arms: Control; Ketamine low-dose
Drug: Ketamine low-dose — Loading: 0.5 mg/Kg Infusion: 5 mcg/kg/min
  Arms: Control; Ketamine high-dose

SUMMARY:
The purpose of this research is to evaluate the effectiveness of ketamine as an analgesic adjuvant in decreasing the narcotic (opioids) analgesics during surgery, on pain management and on the later recovery after surgery in patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
Adjuvant is a drug that has few or no pharmacological effects by itself, but may increase the effectiveness or strength of other drugs when given at the same time.

ELIGIBILITY:
Inclusion Criteria

1. Patients scheduled to undergo small and/or large partial bowel resection via laparotomy or laparoscopy
2. Willingness and ability to sign an informed consent document
3. No allergies to anesthetic or analgesic medications
4. 18 - 80 years of age
5. American Society of Anesthesiologists (ASA) Class I - III adults of either sex

Exclusion Criteria

1. Inability to comprehend the pain assessment tools
2. Patients with known allergy, hypersensitivity or contraindications to anesthetic or analgesic medications
3. Patients with clinically-significant heart disease including arrhythmias and significant hypertension, brain aneurysms, prior history of cerebral vascular accident (CVA), or chronic renal insufficiency
4. Prior abdominal surgery
5. History of abdominal carcinomatosis
6. History of radiation enteritis;
7. Patients with history of hepatic, renal, cardiac failure, organ transplant, or diabetes
8. Patients with seizures
9. Morbid obesity (body mass index >40)
10. Pregnant or lactating women
11. Subjects with a history of alcohol or drug abuse within the past 3 months
12. Any other conditions or use of any medication which may interfere with the conduct of the study
13. Prophylactic Nasogastric Tube (NGT) use
14. Individuals with significant manic disorders including: schizophrenia, or bipolar disorder or psychosis
15. Individuals with asthma and/or thyroid diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD PhD, Principal Investigator — Cedars-Sinai Medical Center; Roya Yumul, MD., PhD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose
Started | 6 | 8 | 7
Completed | 6 | 8 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose | Total
Number analyzed (Participants) | 6 | 8 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (21) | 46 (24) | 58 (12) | 48 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 13
  Male | 3 | 2 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 5 | 7 | 6 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Opioid Consumption
Description: Perioperative use of opioid consumption at Post Anesthesia Care Unit (PACU) Data obtained from patient charts
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose
Number analyzed (Participants) | 6 | 8 | 7
participants | 4 | 5 | 2

2. Secondary Outcome: Postoperative Pain
Description: Postoperative pain was measured at PACU using a Verbal Rating Scale (VRS) from 0 to 10 with 0 representing "no pain" and 10 "very much pain.
Time Frame: one day
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose
Number analyzed (Participants) | 6 | 8 | 7
Score on scale | 5.7 (4.6) | 5.3 (4.6) | 1 (2.2)

3. Secondary Outcome: Participants With Nausea and Vomiting at PACU
Description: Postoperative nausea and vomiting at PACU Participants experiencing nausea and/or vomiting.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose
Number analyzed (Participants) | 6 | 8 | 7
Participants | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Control | Ketamine Low-dose | Ketamine High-dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No